CLINICAL TRIAL: NCT03765463
Title: Extinction Learning in Youth With Tourette Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00195059
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Tourette Syndrome in Children; Tourette Syndrome in Adolescence; Habit Reversal Training; Tic
Keywords: Extinction learning; Behavior Therapy; Tourette's Disorder; Habit Reversal Training; Comprehensive Behavioral Intervention for Tics
MeSH Terms: conditions — Tics; Tourette Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Habit Reversal Training (Experimental): Habit Reversal Training (HRT) is a multi-component evidence-based treatment for tics. It will be delivered over 4 two-hour sessions in an intensive format.
  Interventions: Behavioral: Habit Reversal Training

INTERVENTIONS:
Behavioral: Habit Reversal Training — 4 sessions of habit reversal training

SUMMARY:
Aversive sensory phenomena such as premonitory urges play a central role in the behavioral treatment model of tics. Extinction learning and extinction recall are learning processes implicated within this model, but have not been directly evaluated in youth with Tourette syndrome (TS). This study examines extinction learning and extinction recall in youth with TS using an experimental task. This study will also explore the relationship between extinction processes (i.e., extinction learning and extinction recall) and treatment outcomes with behavior therapy. Findings from this investigation will be used to update the behavioral treatment model, which serves as the basis for evidence-based behavioral interventions.

ELIGIBILITY:
Youth with TS will be eligible for participation if they meet the following inclusion criteria:

* age 8-17 years (inclusive)
* have moderate tic severity or greater as evidenced by a YGTSS Total Tic Score greater than 13 (>9 for youth with motor or vocal tics only)
* have not received more than 4 previous sessions of HRT
* be fluent in English.
* Medication free or on a stable dose of psychiatric medication for 8 weeks prior to enrollment.

Exclusion criteria for youth with TS:

* An inability to complete rating scales
* Attend study visits.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Tic severity as assessed by the Hopkins Motor and Vocal Tic Scale (HM/VTS) | Within 1 week after completion of HRT
  Patient will nominate up to five motor and five vocal tics they deem bothersome on the HM/VTS. Each bothersome tic is then rated by a clinician on the composite two (vocal and motor) 5-point HM/VTS scale ranging from none (0) to severe (4) for the motor as well as vocal tics. The individual tic scores are summed (minimum of 0 and maximum of 40) and averaged together to create an average tic severity score.

SECONDARY OUTCOMES:
Tic severity as assessed by the Yale Global Tic Severity Scale-Revised (YGTSS) | Within 1 week after completion of HRT
  The YGTSS is a clinician-rated semi-structured interview that measures tic symptom severity over the previous week. It consists of 10-items that assess different dimensions of tic severity for motor and vocal tics, which are rated on a 0-5 scale. The YGTSS produces a Total Tic Score (range: 0-50), with higher ratings indicating greater tic severity. The YGTSS has demonstrated treatment sensitivity to pharmacotherapy and behavioral interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F McGuire, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided